CLINICAL TRIAL: NCT05683743
Title: The Incidence, Risk Factors, and Effects of Constipation in Critical Patients: An Observational Cross-sectional Study
Brief Title: The Incidence, Risk Factors, and Effects of Constipation in Critical Patients
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Arzu AKMAN YILMAZ, Asst. Prof, Abant Izzet Baysal University
Other Study IDs: BAIBU-HEM-AAY-001
Record Dates: First submitted 2022-12-16; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Constipation
Keywords: Critical care; Constipation; Intensive care; Nursing
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to investigate the early, late, and total constipation frequency, related factors, and their effects on the hospitalization day, gastric residual volume, vomiting, distension, and diarrhea, the feeding type, white blood cells, and C-Reactive Protein levels, and body temperature.

DETAILED DESCRIPTION:
Constipation is one of the most encountered nursing problems in intensive care unit patients.

Constipation is an important issue, especially in intensive care patients, requiring careful discussion since it has negative effects as well as high incidence and excessive risk factors. Furthermore, untreated constipation in these patients delays enteral feeding prolonging the time of weaning from the mechanical ventilator, which consequently increases the duration of stay in the intensive care unit. Additionally, it involves complications such as distention, nausea-vomiting, an increase in bacterial infection rate, high morbidity, and mortality. Therefore, the definitions, risks, and effects of constipation, especially early and late constipation, in critically ill patients should be determined for evidence-based interventions. However, studies on the subject are limited.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Not abdominal surgery
* Not stoma
* Not constipation during admission
* Not intraperitoneal infection
* Not had a recent colonoscopy -> 5 hospitalization days

Exclusion Criteria:

* Having prolonged constipation and complications (such as decreased bowel sounds, and excessive distension)
* Order for regular laxatives or enemas
* Not meet inclusion criteria during follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data were collected from the Anesthesia and Reanimation Intensive Care Unit in a state hospital of Bolu in 2019. To determine the number of observations in our study, a pilot study was conducted with 20 patients. These patients were also included in the main study. The constipation rate in the intensive care unit was determined as 67% in the pilot study. Considering this ratio, the sample size was calculated using the PASS 11 program. Accordingly, at least 86 patients had to be included in the study keeping a 95% probability and 10% deviation. The sample consisted of 116 patients who were reachable during the study, met the inclusion criteria, and volunteered to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
The frequency of total constipation, early-type constipation and late-type constipation | Through study completion, an average of five months
  During the study, patients in the intensive care unit with no bowel movements for four days were accepted as constipated. The ones without defecation for five days were evaluated in the early type constipation group, while the patients without defecation for six days or more were evaluated in the late-type constipation group.

SECONDARY OUTCOMES:
he duration of stay in the intensive care unit | Through study completion, an average of five months
  the duration of stay in the intensive care unit as days (how many days?)
the amount of gastric residual volume | Through study completion, an avarage of five months
  the amount of gastric residual volume in ml/cc
developing vomiting | Through study completion, an average of five months
  developing vomiting as numbers (how many times?)
Level of white blood cells | Through study completion, an average of five months
  level of white blood cells (WBC) in mcL
body temperature | Through study completion, an average of five months
  body temperature in celsius

CONTACTS AND LOCATIONS:
Overall Officials: Arzu AKMAN YILMAZ, RN, PhD., Principal Investigator — Bolu Izzet Baysal University; Seyma OZDEMIR, RN,MSN., Principal Investigator — Pursaklar State Hospital; Esra OZDEMIR, MD., Principal Investigator — Bolu Izzet Baysal State Hospital
Locations (1):
- Bolu Izzet Baysal State Hospital, Anesthesia Intensive Care Unit, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No